CLINICAL TRIAL: NCT02948062
Title: Early Diagnosis Of Childhood Cerebral Adrenoleukodystrophy
Brief Title: Early Diagnosis Of Childhood Cerebral ALD
Status: Withdrawn | Type: Observational
Why Stopped: Funding unavailable
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2016NTLS155; MT2016-29R (Other: University of Minnesota)
Record Dates: First submitted 2016-10-25; First posted 2016-10-28 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Adrenoleukodystrophy
Keywords: ALD; Newborn Screening
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and cerebral spinal fluid.

SUMMARY:
The goal of this single institution study is to evaluate boys with adrenoleukodystrophy (ALD) diagnosed early in life, and to prospectively monitor them to determine parameters that will facilitate earlier detection of the childhood cerebral form of the disease. These at-risk subjects will be assessed yearly through travel to the University of Minnesota, where plasma and cerebral spinal fluid (CSF) biomarker studies, MRI based imaging and neuropsychological assessments will be performed at the University of Minnesota Masonic Children's Hospital and Clinics. The MRI and lumbar puncture to obtain CSF will be obtained under sedation. In addition, at intervening 6 months intervals information will be obtained remotely, including surveys and MRI's in their home location. Also at that time blood samples will be obtained locally and shipped to the University of Minnesota for study. There is no therapeutic intent in this study.

ELIGIBILITY:
Inclusion Criteria:

* Boys with confirmed adrenoleukodystrophy, as determined by very long chain fatty acid (VLCFA) analysis and/or genotyping. Genotyping is not necessary for diagnosis.
* Between 1 and 5 years of age, inclusive at the time of consent.
* Able to undergo a sedation
* English as primary language of the household, to maximize consistency of the neuropsychological/developmental testing.
* Voluntary written parental/guardian consent

Exclusion Criteria:

* Evidence of cerebral disease at time of enrollment - patients over 3 years of age must have an MRI within 4 months of signing consent to confirm that there is no evidence of cerebral disease
* Inability or unwillingness to travel to the University of Minnesota once a year for the duration of the study
* Evidence of cerebral disease by standard T2/FLAIR MRI. If a subject develops cerebral ALD during the study, they will come off study, as it is anticipated that they would be considered for transplantation.

Ages: 1 Year to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: While this study will be registered with clinicaltrials.gov, no specific patient recruitment materials will be utilized. However, various Foundations and Patient Groups will be contacted. In addition, we will work with providers, neurologists, genetic counselors, etc. in the areas where newborn screening is taking place. We will also be available for families and providers at other institutions where a diagnosis may be made.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
ALD Early Evaluation | 5 years
  To evaluate boys with adrenoleukodystrophy (ALD) diagnosed early in life, and to prospectively determine factors that have a high correlation with the emergence of cerebral ALD.

SECONDARY OUTCOMES:
Emergence of cerebral disease through imaging | 5 years
  The ability to discern the emergence of cerebral disease through imaging prior to the onset of classic T2 imaging. This will include diffusion tensor imaging (DTI), T1 and T2 rho, RAFF and spectroscopy, in addition to the standard MRI evaluations including gadolinium enhancement.
Biomarker Study: Inflammation Markers | 5 years
  Markers of inflammation (chitotriosidase, lipidomics including arachidonic acid metabolites and inflammatory cytokines).
Biomarker Study: Oxidative Stress | 5 years
  Determinations of oxidative stress (including but not limited to total and reduced/oxidized glutathione and 4-hydroxynonenal, or 4-HNE).
Biomarker Study: Immunologic Activation | 5 years
Neuropsychology testing | 5 years
  Extensive neuropsychology testing, including assessments of verbal comprehension, perceptual reasoning, working memory and processing speed.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States